CLINICAL TRIAL: NCT07107048
Title: Clinical Prospective Randomized Trial to Evaluate the Non-inferiority of Left Bundle Branch Area Pacing vs Cardiac Resynchronization Therapy With ECG Guided AV Optimization (DA VINCI STUDY)
Brief Title: Clinical Prospective ranDomized Trial to Evaluate the Non-inferiority of Left Bundle Branch Area Pacing Vs Cardiac ResynchronIzatioN Therapy With ECG guIded AV Optimization
Acronym: DA VINCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leonardo Calò, MD (Other)
Collaborators: National association Cardiovascular innovation (Unknown)
Responsible Party: Sponsor-Investigator, Leonardo Calò, MD, Prof., Policlinico Casilino ASL RMB
Organization: Policlinico Casilino ASL RMB (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v1 7jul25
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
Keywords: lbbap; crt
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked | interventions — Defibrillators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBAP (Experimental): Patients undergoing left bundle branch area pacing (LBBAP) implantation
  Interventions: Device: Pacemaker and defibrillator
- CRT Biv (Active Comparator): Patients undergoing cardiac resynchronization therapy (CRT) with biventricular pacing
  Interventions: Device: Pacemaker and defibrillator

INTERVENTIONS:
Device: Pacemaker and defibrillator — Patients will be randomly assigned at enrollment (1:1) to undergo either LBBAP or CRT with biventricular stimulation. The devices implanted maybe defibrillators or pacemekers.

SUMMARY:
Cardiac resynchronization therapy is the gold standard therapy for patients with advanced HF left ventricle dysfunction and large QRS.

Recently left bundle branch area pacing (LBBAP) or left bundle optimized cardiac resynchronization therapy has been proposed as a rescue therapy for failed or unsuccessful CRT. LBBAP has been also proposed as a physiological pacing modality for patient who need permanent ventricular pacing as an alternative to conventional right ventricular pacing.

Several observational studies have demonstrated the feasibility of this technique due to an ease procedure, stable and appropriate electrical measurements and clinical benefit in terms of patients outcomes.

Furthermore, It is well known that an optimized AV delay (AVD) can improve clinical outcomes preserving a physiological diastolic function.

In clinical practice several different AVD optimization methods have been developed in the last few years.

The majority of them use the intracardiac electrograms during the implant procedure to evaluate QRS duration and AV delay or at follow-up through echocardiographic measurements.

Aim of our pilot project is to assess the non-inferiority of Left Bundle Branch Area Pacing vs Cardiac Resynchronization Therapy with ECG/Echo guided AV optimization.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy is the gold standard therapy for patients with advanced HF left ventricle dysfunction and large QRS.

Recently left bundle branch area pacing (LBBAP) or left bundle optimized cardiac resynchronization therapy has been proposed as a rescue therapy for failed or unsuccessful CRT. LBBAP has been also proposed as a physiological pacing modality for patient who need permanent ventricular pacing as an alternative to conventional right ventricular pacing.

Several observational studies have demonstrated the feasibility of this technique due to an ease procedure, stable and appropriate electrical measurements and clinical benefit in terms of patients outcomes.

Furthermore, LBBAP provides a fast activation of the left ventricle and has shown to maintain electrical synchrony shortening the QRS and providing the correction of left bundle branch block (LBBB) by pacing beyond the block.

Despite of that, it is common to find right bundle branch block (RBBB) at the electrocardiography (ECG) that represents a delay in the RV activation and interventricular dissynchrony.

This finding in patients with heart failure may worsen their conditions as shown in literature.

RBBB may be minimized by the resynchronization of right ventricle and left ventricle with an adequate time sequence or by the correct optimization of the atrioventricular delay for both CRT and LBBAP in order to enable fusion with intrinsic RV conduction in patients without a complete AV block.

It is well known that an optimized AV delay (AVD) can improve clinical outcomes preserving a physiological diastolic function.

In clinical practice several different AVD optimization methods have been developed in the last few years.

The majority of them use the intracardiac electrograms during the implant procedure to evaluate QRS duration and AV delay or at follow-up through echocardiographic measurements.

Among all the echocardiographic modalities, the mitral inflow velocity time integral (VTI) is a surrogate for LV filling volume assuming a constant mitral valve area. Mitral inflow is dependent on timing of both left atrial and left ventricular systole, and interatrial and interventricular conduction delays will affect optimal timing of ventricular pacing.

Aim of our pilot project is to assess the non-inferiority of Left Bundle Branch Area Pacing vs Cardiac Resynchronization Therapy with ECG/Echo guided AV optimization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indications of cardiac resynchronization therapy
* Patients with Left Branch Block (LBBB) (2021 ESC/REVERSE. Glickson et al _EHJ 2021):
* Patients over 18 years of age.

Exclusion Criteria:

* • Women who are pregnant, lactating, or plan to become pregnant during the trial.

  * 3rd degree AV Block
  * Participants with angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary, intervention in the next three (3) months.
  * Enzyme-positive myocardial infarction within the past three (3) months prior to enrollment.
  * Coronary artery bypass graft surgery or percutaneous coronary intervention (balloon and/or stent angioplasty) within the past three (3) months prior to enrollment.
  * Reversible non-ischemic cardiomyopathy (e.g., acute viral myocarditis).
  * Participants with Chagas disease, cardiac sarcoidosis or amyloidosis.
  * Expected to receive left ventricular assist device or heart transplantation within 6 months.
  * Participants with severe valvular disease (e.g., aortic stenosis).
  * Have a life expectancy of less than 12 months.
  * Participants with irreversible brain damage from preexisting cerebral disease.
  * Participants with a contrast dye allergy unable or unwilling to undergo pretreatment with steroids and/or diphenhydramine.
  * Long-lasting or permanent atrial fibrillation
  * Participants participating in any other interventional cardiovascular clinical trial.
  * Participants who would be unable to return for follow-up visits due to the distance from the clinic.
  * Participants who do not anticipate being a resident of the area for the scheduled duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 194 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
CRT response | 6 months
  CRT RESPONSE WILL BE DEFINED:
  * Freedom from HF Hospitalizations
  * Freedom from Cardiac Death
  * Reverse remodeling: ≥15% relative reduction in left ventricular end-systolic volume

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Casilino, Rome, Italy

IPD SHARING:
Plan to Share IPD: No